CLINICAL TRIAL: NCT04944160
Title: Impact of the Covid-19 Pandemic on the Epidemiology of Respiratory Syncytial Virus
Brief Title: Impact of the Covid-19 on Respiratory Syncytial Virus (RSV) Epidemic
Acronym: IPCoVRS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 502
Record Dates: First submitted 2021-06-28; First posted 2021-06-29 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2021-06

CONDITIONS: RSV Infection
Keywords: bronchiolitis; Asthma; Pneumonia
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Bronchiolitis; Asthma; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre Covid-19 cohort: Children hospitalized in the Pediatric Department of the " Hôpital Femme Mère Enfant ", Lyon, France with a reverse transcriptase - polymerase chain reaction (RT-PCR) positive for Respiratory Syncytial Virus (RSV) during the 2019-2020 winter epidemic
  Interventions: Other: Medical records analysis; Other: Comparison of cohorts
- Post Covid-19 cohort: Children hospitalized in the Pediatric Department of the " Hôpital Femme Mère Enfant ", Lyon, France with a reverse transcriptase - polymerase chain reaction (RT-PCR) positive for Respiratory Syncytial Virus (RSV) during the 2020-2021 winter epidemic
  Interventions: Other: Medical records analysis; Other: Comparison of cohorts

INTERVENTIONS:
Other: Medical records analysis — To review of medical records to describe diagnosis and severity of the disease.
Other: Comparison of cohorts — To compare pre and post Covid-19 epidemics in terms of numbers of admissions, and proportion of severe disease.
  Other Names: Epidemiology

SUMMARY:
The magnitude of seasonal Respiratory Syncytial Virus (RSV) epidemics brings each year new logistical challenges for the hospitalization of young infants with bronchiolitis that overwhelm hospital capacities and lead to specific winter plans with deprogramming and mobilization of human and logistical resources. The Covid-19 pandemic has changed the way winter epidemics are presented. For example, the seasonal RSV epidemic was shifted by several months in Lyon, with an impression of a lower incidence of hospitalized cases, with a population of older children and with fewer signs of clinical severity. This is largely attributable to the widespread use of barrier gestures and social distancing measures, known as "Non-Pharmacological Interventions" (NPI). Given the magnitude of the reduction of the RSV epidemic, it is legitimate to analyze the benefits of NPIs to draw lessons for maintaining preventive measures around RSV-vulnerable populations; moreover, new preventive pharmacological interventions are soon to be marketed, whether they are particularly refined and long half-life anti-RSV monoclonal antibodies, RSV vaccines for mothers or for newborns and infants. In this perspective, it is crucial to properly define the populations at risk of severe disease to establish a legitimate hierarchy in the implementation of different preventive strategies. The study of the RSV epidemic is a high potential model because of the convergence of epidemiological, virological, and pharmacological knowledge. However, the study of the impact of the pandemic on the epidemiology of rhinovirus also seems promising because, for reasons unknown to date, it seems that the pandemic did not have the same reducing impact on the rhinovirus epidemic; in the latter case, the interest is to confirm the resistance of this virus and to look for more fundamental explanations, for example, on viral interactions.

ELIGIBILITY:
Inclusion Criteria:

* • Child hospitalized at " Hôpital Femme Mère Enfant ", Lyon, France

  * Polymerase Chain Reaction (PCR) positive at Respiratory Syncytial Virus (RSV)

Exclusion Criteria:

* • Parent's refusal to participate

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Child hospitalized at " Hôpital Femme Mère Enfant ", Lyon, France with viral respiratory infection.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Reduction of the number of children hospitalized for a RSV-infection during pre and post-Covid-19 pandemic RSV-winter-epidemic. | 2019-2020-winter-epidemic and 2020-2021-winter-epidemic are assessed during June and July, 2021.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupement Hospitalier EST - Hospices Civils de Lyon, Bron, France

REFERENCES:
- [Derived] Casalegno JS, Ploin D, Cantais A, Masson E, Bard E, Valette M, Fanget R, Targe SC, Myar-Dury AF, Doret-Dion M, Massoud M, Queromes G, Vanhems P, Claris O, Butin M, Pillet S, Ader F, Bin S, Gaymard A, Lina B, Morfin F; VRS study group in Lyon; Javouhey E, Gillet Y. Characteristics of the delayed respiratory syncytial virus epidemic, 2020/2021, Rhone Loire, France. Euro Surveill. 2021 Jul;26(29):2100630. doi: 10.2807/1560-7917.ES.2021.26.29.2100630. PMID 34296674